CLINICAL TRIAL: NCT04206514
Title: Strengthening Patient-Centered Accessibility, Respect, and Quality of Care for Post Abortion Care Through Peer and Nurse Based Phone Support
Brief Title: Improving Person Centered Care for Post Abortion Patients in Kenya
Acronym: SPARQ_PACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Innovations for Poverty Action (Other); Marie Stopes International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-18008_Kenya Abortion
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Reproductive Health
Keywords: post abortion; person-centered care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer Counselor (Experimental): Participants receive personalized text messages and phone calls from a peer counselor- a women who had an abortion and was trained in post abortion care and PCC
  Interventions: Behavioral: Person Centered Care - Post Abortion Support
- Nurse (Experimental): Participants receive personalized text messages and phone calls from a nurse trained in post abortion care and PCC
  Interventions: Behavioral: Person Centered Care - Post Abortion Support
- control (No Intervention): Participants receive the standard of care for post-abortion patients in Kenya.

INTERVENTIONS:
Behavioral: Person Centered Care - Post Abortion Support — Post abortion phone based support
  Arms: Nurse; Peer Counselor

SUMMARY:
The purpose of this study is to understand the effect of a phone based post-abortion intervention on the experience of post-abortion care.

DETAILED DESCRIPTION:
This study evaluates whether personalized text messages and phone calls to post abortion women can improve post abortion person-centered care, perceived social support, post-abortion family planning, and reduce perceptions of social stigma and stress. Women were randomized to one of three study arms: personalized communication with a peer counselor or nurse who received person-centered care (PCC) training, or a control arm where participants received the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age
* Had an Safe Abortion (SA)/Post Abortion Care (PAC) procedure at one of six private clinics that day
* Has her own cellphone that is WhatsApp compatible and will have access to this phone for the next four weeks
* Willing to receive receive short message service (SMS) messages and phone calls from an Marie Stopes Kenya (MSK) or Innovation for Poverty Action (IPA) professional
* Able to communicate in English and/or Swahili
* Willing and able to comprehend and give informed consent
* Willing to participate in a baseline survey immediately after providing consent
* Willing to be followed up by phone at two weeks and four weeks post procedure for a 15-minute survey at each time-point
* Has not already participated in this study

Exclusion Criteria:

* Is not a women of reproductive age
* Did not have an SA/PAC procedure at one of six private clinics that day
* Does not have her own cellphone that is WhatsApp compatible and will have access to this phone for the next four weeks
* Is not willing to SMS messages and phone calls from an MSK/IPA professional
* Is not able to communicate in English and/or Swahili
* Is not willing or is not able to comprehend and give informed consent
* Is not willing to participate in a baseline survey immediately after providing consent
* Is not willing to be followed up by phone at two weeks and four weeks post procedure for a 15-minute survey at each time-point
* Has already participated in this study

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 371 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Person-Centered Abortion Scale Score | baseline
  Survey conducted with women: self-report of experiences of PCC. Possible range 0-100; higher the score, better the experience
Person-Centered Abortion Scale Score | 2 weeks post-procedure
  Survey conducted with women: self-report of experiences of PCC. Possible range 0-100; higher the score, better the experience
Person-Centered Abortion Scale Score | 4 weeks post-procedure
  Survey conducted with women: self-report of experiences of PCC. Possible range 0-100; higher the score, better the experience

SECONDARY OUTCOMES:
Post abortion family planning counseling | baseline
  Self-report if women received counseling on family planning (Yes/No)
Post-abortion family planning uptake | baseline
  Self-report of uptake of family planning (Yes/No/Refused to answer)
Perceived social support | baseline
  Medical Outcomes Study-Social Support 15-item Scale (MOS-SSS): 18-90 where higher scores indicate greater social support
Perceived abortion stigma | baseline
  The Individual Level Abortion Stigma Scale (ILAS Scale) Abbreviated 3-item Scale: 0-9 where higher scores indicate greater worry about stigma
Mental Health | baseline
  Mental Health Inventory (MHI-5) scale; 0-100 with higher scores indicating better mental health
Post-abortion family planning uptake | 2 weeks post-procedure
  self-report of uptake of family planning (Yes/No/Refused to answer)
Mental Health | 2-weeks post procedure
  Mental Health Inventory (MHI-5) scale; 0-100 with higher scores indicating better mental health
Post-abortion family planning uptake | 4 weeks post-procedure
  self-report of uptake of family planning (Yes/No/Refused to answer)
Perceived social support | 4 weeks post-procedure
  Medical Outcomes Study-Social Support 15-item Scale (MOS-SSS): 18-90 where higher scores indicate greater social support
Perceived abortion stigma | 4 weeks post procedure
  The Individual Level Abortion Stigma Scale (ILAS Scale) Abbreviated 3-item Scale: 0-9 where higher scores indicate greater worry about stigma

CONTACTS AND LOCATIONS:
Overall Officials: May Sudhinaraset, PhD, Principal Investigator — University of California, San Francisco/University of California, Los Angeles
Locations (1):
- Marie Stopes International Kenya, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allison S, Bauermeister JA, Bull S, Lightfoot M, Mustanski B, Shegog R, Levine D. The intersection of youth, technology, and new media with sexual health: moving the research agenda forward. J Adolesc Health. 2012 Sep;51(3):207-12. doi: 10.1016/j.jadohealth.2012.06.012. PMID 22921129
- [Background] Amirkhanian YA, Kelly JA, Kabakchieva E, McAuliffe TL, Vassileva S. Evaluation of a social network HIV prevention intervention program for young men who have sex with men in Russia and Bulgaria. AIDS Educ Prev. 2003 Jun;15(3):205-20. doi: 10.1521/aeap.15.4.205.23832. PMID 12866833
- [Background] Brookman-Amissah E, Moyo JB. Abortion law reform in sub-Saharan Africa: no turning back. Reprod Health Matters. 2004 Nov;12(24 Suppl):227-34. doi: 10.1016/s0968-8080(04)24026-5. PMID 15938178
- [Background] Bull SS, Levine DK, Black SR, Schmiege SJ, Santelli J. Social media-delivered sexual health intervention: a cluster randomized controlled trial. Am J Prev Med. 2012 Nov;43(5):467-74. doi: 10.1016/j.amepre.2012.07.022. PMID 23079168
- [Background] Ceylan A, Ertem M, Saka G, Akdeniz N. Post abortion family planning counseling as a tool to increase contraception use. BMC Public Health. 2009 Jan 15;9:20. doi: 10.1186/1471-2458-9-20. PMID 19146657
- [Background] Charles VE, Polis CB, Sridhara SK, Blum RW. Abortion and long-term mental health outcomes: a systematic review of the evidence. Contraception. 2008 Dec;78(6):436-50. doi: 10.1016/j.contraception.2008.07.005. Epub 2008 Sep 23. PMID 19014789
- [Background] Cuijpers P. Effective ingredients of school-based drug prevention programs. A systematic review. Addict Behav. 2002 Nov-Dec;27(6):1009-23. doi: 10.1016/s0306-4603(02)00295-2. PMID 12369469
- [Background] Desai M, Phillips-Howard PA, Odhiambo FO, Katana A, Ouma P, Hamel MJ, Omoto J, Macharia S, van Eijk A, Ogwang S, Slutsker L, Laserson KF. An analysis of pregnancy-related mortality in the KEMRI/CDC health and demographic surveillance system in western Kenya. PLoS One. 2013 Jul 16;8(7):e68733. doi: 10.1371/journal.pone.0068733. Print 2013. PMID 23874741
- [Background] Evens E, Otieno-Masaba R, Eichleay M, McCarraher D, Hainsworth G, Lane C, Makumi M, Onduso P. Post-abortion care services for youth and adult clients in Kenya: a comparison of services, client satisfaction and provider attitudes. J Biosoc Sci. 2014 Jan;46(1):1-15. doi: 10.1017/S0021932013000230. Epub 2013 Jun 10. PMID 23745828
- [Background] Harris GE, Larsen D. HIV peer counseling and the development of hope: perspectives from peer counselors and peer counseling recipients. AIDS Patient Care STDS. 2007 Nov;21(11):843-60. doi: 10.1089/apc.2006.0207. PMID 18240894
- [Background] Ikamari L, Izugbara C, Ochako R. Prevalence and determinants of unintended pregnancy among women in Nairobi, Kenya. BMC Pregnancy Childbirth. 2013 Mar 19;13:69. doi: 10.1186/1471-2393-13-69. PMID 23510090
- [Background] Kelly JA, Murphy DA, Sikkema KJ, McAuliffe TL, Roffman RA, Solomon LJ, Winett RA, Kalichman SC. Randomised, controlled, community-level HIV-prevention intervention for sexual-risk behaviour among homosexual men in US cities. Community HIV Prevention Research Collaborative. Lancet. 1997 Nov 22;350(9090):1500-5. doi: 10.1016/s0140-6736(97)07439-4. PMID 9388397
- [Background] Latkin CA, Sherman S, Knowlton A. HIV prevention among drug users: outcome of a network-oriented peer outreach intervention. Health Psychol. 2003 Jul;22(4):332-9. doi: 10.1037/0278-6133.22.4.332. PMID 12940388
- [Background] Lightfoot M, Comulada WS, Stover G. Computerized HIV preventive intervention for adolescents: indications of efficacy. Am J Public Health. 2007 Jun;97(6):1027-30. doi: 10.2105/AJPH.2005.072652. Epub 2006 May 2. PMID 16670219
- [Background] Magadi MA. Unplanned childbearing in Kenya: the socio-demographic correlates and the extent of repeatability among women. Soc Sci Med. 2003 Jan;56(1):167-78. doi: 10.1016/s0277-9536(02)00018-7. PMID 12435559
- [Background] Mellanby AR, Newcombe RG, Rees J, Tripp JH. A comparative study of peer-led and adult-led school sex education. Health Educ Res. 2001 Aug;16(4):481-92. doi: 10.1093/her/16.4.481. PMID 11525394
- [Background] Mohamed SF, Izugbara C, Moore AM, Mutua M, Kimani-Murage EW, Ziraba AK, Bankole A, Singh SD, Egesa C. The estimated incidence of induced abortion in Kenya: a cross-sectional study. BMC Pregnancy Childbirth. 2015 Aug 21;15:185. doi: 10.1186/s12884-015-0621-1. PMID 26294220
- [Background] Oyieke JB, Obore S, Kigondu CS. Millennium development goal 5: a review of maternal mortality at the Kenyatta National Hospital, Nairobi. East Afr Med J. 2006 Jan;83(1):4-9. doi: 10.4314/eamj.v83i1.9345. PMID 16642744
- [Background] Pulerwitz J, Michaelis A, Verma R, Weiss E. Addressing gender dynamics and engaging men in HIV programs: lessons learned from Horizons research. Public Health Rep. 2010 Mar-Apr;125(2):282-92. doi: 10.1177/003335491012500219. PMID 20297757
- [Background] Steinberg JR, Tschann JM, Furgerson D, Harper CC. Psychosocial factors and pre-abortion psychological health: The significance of stigma. Soc Sci Med. 2016 Feb;150:67-75. doi: 10.1016/j.socscimed.2015.12.007. Epub 2015 Dec 12. PMID 26735332
- [Background] Teti M, Rubinstein S, Lloyd L, Aaron E, Merron-Brainerd J, Spencer S, Ricksecker A, Gold M. The Protect and Respect program: a sexual risk reduction intervention for women living with HIV/AIDS. AIDS Behav. 2007 Sep;11(5 Suppl):S106-16. doi: 10.1007/s10461-007-9275-y. Epub 2007 Jun 29. PMID 17605102
- [Background] Turner G, Shepherd J. A method in search of a theory: peer education and health promotion. Health Educ Res. 1999 Apr;14(2):235-47. doi: 10.1093/her/14.2.235. PMID 10387503
- [Background] Upadhyay UD, Cockrill K, Freedman LR. Informing abortion counseling: an examination of evidence-based practices used in emotional care for other stigmatized and sensitive health issues. Patient Educ Couns. 2010 Dec;81(3):415-21. doi: 10.1016/j.pec.2010.08.026. PMID 20926226
- [Background] Yegon EK, Kabanya PM, Echoka E, Osur J. Understanding abortion-related stigma and incidence of unsafe abortion: experiences from community members in Machakos and Trans Nzoia counties Kenya. Pan Afr Med J. 2016 Jul 20;24:258. doi: 10.11604/pamj.2016.24.258.7567. eCollection 2016. PMID 27800111
- [Background] Ziraba AK, Madise N, Mills S, Kyobutungi C, Ezeh A. Maternal mortality in the informal settlements of Nairobi city: what do we know? Reprod Health. 2009 Apr 22;6:6. doi: 10.1186/1742-4755-6-6. PMID 19386134